CLINICAL TRIAL: NCT04790604
Title: Enhancing Community Health Through Patient Navigation, Advocacy and Social Support (ENCOMPASS): Expansion Study A, A Randomized Controlled Trial With Waitlist Control
Brief Title: ENCOMPASS: Expansion Study A, RCT
Acronym: ENCOMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REB19-1766
Record Dates: First submitted 2021-01-13; First posted 2021-03-10 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2; Chronic Kidney Diseases; Ischemic Heart Disease; Congestive Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma
Keywords: Chronic Disease; Health Navigation; Health Navigator
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Myocardial Ischemia; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Chronic Disease

STUDY DESIGN:
Intervention Model Description: The ENCOMPASS study will evaluate the effectiveness of a community health navigator program using a two-armed, pragmatic, randomized waitlist-controlled trial. The intervention arm will receive the CHN program for six months. The waitlist control arm will have a six month waiting period followed by six months of CHN program. This study will employ patient-level block randomization. Research staff will be blinded to block size. In the case where participants live together in the same residence, they will be randomly assigned to the same study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Community health navigator program for six months.
  Interventions: Behavioral: Community Health Navigator Program
- Control (Other): Waitlist control: six-month waiting period followed by six months of community health navigator program.
  Interventions: Behavioral: Community Health Navigator Program

INTERVENTIONS:
Behavioral: Community Health Navigator Program — Patients will be matched to a community health navigator (CHN) who will conduct a needs assessment to determine the frequency of meetings. A CHN may perform any of the following: providing information to a patient's health care provider, translation, advocating for the patient, connecting the patient with resources (e.g., social, financial, insurance), helping patients set health-related goals, facilitating health care referrals and appointments, and monitoring appointments. These activities may require the CHN to be physically present at appointments or have direct contact with the patient's health care provider. Goal setting and support will be provided in-person or over the telephone using motivational interviewing principles.
  Other Names: ENCOMPASS Program

SUMMARY:
Some patients living with multiple long-term health conditions have difficulty accessing the services they need, despite available primary care and community resources. Patient navigation programs may help those with complex health conditions to improve their care and outcomes. Community health navigators (CHNs) are community members who help guide patients through the health care system. CHNs are not health professionals like a doctor or nurse, but they are specially trained to help patients get the most out of their health care and connect them to resources. The ENCOMPASS program of research evaluates a patient navigation program that connects patients living with long-term health conditions to CHNs. To understand if the CHN program can be scaled to a provincial level, the ENCOMPASS program of research is expanding to select primary care settings across Alberta. This study implements and evaluates the CHN program at Edmonton Oliver Primary Care Network in Edmonton, Alberta, Canada.

DETAILED DESCRIPTION:
Community Health Navigators (CHNs) are defined as community health workers that provide patient navigation. Based on evidence to date, CHNs for chronic disease management are likely to beneficially impact patient experience, clinical outcomes and costs; however, contextual evidence is lacking given that most studies to date have been conducted in the United States. In Canada, patient navigation programs currently exist in only a few settings (primarily cancer treatment and transitional care), with few navigation programs implemented in chronic disease care.

The ENCOMPASS program of research was initiated in 2016, when researchers with the University of Calgary's Interdisciplinary Chronic Disease Collaboration partnered with Mosaic Primary Care Network (PCN) to develop, implement and evaluate a community health navigation program for patients with multiple chronic conditions. The program was based on a systematic literature review and refined in consultation with key stakeholders. A cluster-randomized controlled trial is currently ongoing with Mosaic PCN to determine the impact of the program on acute care use, patient-reported outcomes and experience, and disease-specific clinical outcomes (NCT03077386).

Alberta Primary Care Networks (PCNs) are comprised of groups of family physicians and other health care professionals working together to provide comprehensive patient care to Albertans. To understand if the community health navigation program can be feasibly scaled and spread to PCNs across Alberta, we are expanding research to examine and evaluate community health navigation program implementation to other geographic areas and populations. This study expands the ENCOMPASS program of research to Edmonton Oliver PCN, which represents over 170 physician members and serves approximately 131,000 patients. The current study employs the RE-AIM framework (reach, effectiveness, adoption, implementation, and maintenance) to examine the scalability of the community health navigation program.

The objectives of this study are to (1) assess the impact of the intervention on the target population and health system (effectiveness); (2) explore the feasibility and appropriateness of practical intervention scale-up (reach, adoption, implementation, and maintenance), and (3) identify the required resources and infrastructure necessary to maintain and scale the intervention provincially.

The effectiveness of the community health navigator program will be studied using a two-armed, pragmatic, randomized waitlist-controlled trial. This study will employ patient-level block randomization with research staff blinded to block size. Randomization will be concealed and computer-generated. Primary outcomes will be assessed using administrative health data. Secondary outcomes will be measured using a patient health survey administered by a research assistant at baseline, 6 months, and 12 months. A concurrent qualitative study will provide contextual information on the effectiveness of the community health navigator program from patient, provider, and CHN perspectives. Process evaluation metrics and interviews with program stakeholders will inform the feasibility and sustainability of the community health navigator program in Alberta PCNs.

ELIGIBILITY:
Inclusion Criteria:

* Poorly controlled hypertension (most recent systolic blood pressure > 160 mmHg or labile);
* Poorly controlled diabetes (A1C > 9% on at least one occasion within the past year or labile);
* Stage 3b or greater chronic kidney disease (estimated glomerular filtration rate < 45 mL/min/1.73m2 in past year);
* Established ischemic heart disease (at least one instance of a physician billing diagnosis with a relevant International Classification of Diseases, 9th Edition [ICD-9] code recorded in electronic medical record (EMR), or known to health care team);
* Congestive heart failure (at least one instance of a physician billing diagnosis with a relevant ICD-9 code recorded in EMR, or known to health care team);
* Chronic obstructive pulmonary disease OR Asthma with at least two visits in the past year (at least 2 instances of a physician billing diagnosis with a relevant ICD-9 code, or known to health care team).

Exclusion Criteria:

* Patient unable to provide informed consent;
* Patient residing in long-term care facility;
* Health care provider discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Acute care service use | Up to 36 months
  Rate of emergency department visits and hospital admissions based on administrative health data.

SECONDARY OUTCOMES:
Health-related quality of life | Up to 12 months
  EuroQol EQ-5D-5L.
Patient experience of care | Up to 12 months
  11-item modified Patient Assessment of Chronic Illness Care (PACIC).
Patient activation | Up to 12 months
  10-item Patient Activation Measure (PAM-10), score and level.
Anxiety symptoms | Up to 12 months
  7-item Generalized Anxiety Disorder (GAD-7).
Depressive symptoms | Up to 12 months
  9-item Patient Health Questionnaire (PHQ-9).
Perceived social support | Up to 12 months
  8-item modified Medical Outcomes Study Social Support Survey (mMOS-SS).
Health literacy | Up to 12 months
  3-item Brief Screening Questions for Health Literacy.
General self-rated health | Up to 12 months
  1-item Self-Rated Health (SRH).
Household food security | Up to 12 months
  6-item Household Food Security Survey Module (HFSSM).
Smoking status | Up to 12 months
  Self-reported smoking status.
Weight | Up to 12 months
  Change in self-reported weight in kilograms or pounds.
Disease-specific intermediate health outcomes: Diabetes | Up to 24 months
  Change in mean glycosylated hemoglobin (A1C) based on laboratory data.
Disease-specific intermediate health outcomes: Hypertension | Up to 12 months
  Change in systolic blood pressure (SBP) in mmHg based on primary data collection.
Disease-specific intermediate health outcomes: Heart failure | Up to 24 months
  Episodes of acutely decompensated heart failure based on administrative health data.
Disease-specific intermediate health outcomes: COPD/asthma | Up to 24 months
  Exacerbations based on administrative health data.
Disease-specific intermediate health outcomes: Ischemic heart disease, chronic kidney disease, diabetes | Up to 24 months
  Appropriate use of a statin where indicated based on pharmaceutical information network (PIN) dispensation data.
Patient experience | Up to 12 months
  Based on semi-structured interviews.
Provider satisfaction | Up to 12 months
  Based on semi-structured interviews.
Continuity of care | Up to 24 months
  Provider attachment based on Usual Provider of Care (UPC) Index in Alberta practitioners claims file.
Primary Care Network (PCN) multidisciplinary team access | Up to 24 months
  Number of visits to multidisciplinary health team members based on PCN records.
Program costs | Up to 24 months
  Administrative, training, and operational costs of program.
Physician costs | Up to 24 months
  Physician claims based on physician claims files.
Acute care costs | Up to 24 months
  Hospital admission and emergency department visit costs based on administrative health data.
All-cause mortality | Up to 24 months
  All-cause mortality rate based on administrative data.
Medication adherence | Up to 24 months
  ≥80% of days covered for medications in Care Plan based on pharmaceutical information network (PIN) dispensation data.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry A McBrien, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- Edmonton Oliver Primary Care Network, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehmann U, Sanders, D. Community health workers: What do we know about them? The state of the evidence on programmes, activities, costs an impact on health outcomes of Using community health workers. Geneva: World Health Organization. 2007.
- [Background] Najafizada SA, Bourgeault IL, Labonte R, Packer C, Torres S. Community health workers in Canada and other high-income countries: A scoping review and research gaps. Can J Public Health. 2015 Mar 12;106(3):e157-64. doi: 10.17269/cjph.106.4747. PMID 26125243
- [Background] Addressing chronic disease through community health workers: A policy and systems-level approach. Centers for Disease Control and Prevention. 2015.
- [Background] Kangovi S, Grande D, Trinh-Shevrin C. From rhetoric to reality--community health workers in post-reform U.S. health care. N Engl J Med. 2015 Jun 11;372(24):2277-9. doi: 10.1056/NEJMp1502569. No abstract available. PMID 26061832
- [Background] Burns ME, Galbraith AA, Ross-Degnan D, Balaban RB. Feasibility and evaluation of a pilot community health worker intervention to reduce hospital readmissions. Int J Qual Health Care. 2014 Aug;26(4):358-65. doi: 10.1093/intqhc/mzu046. Epub 2014 Apr 16. PMID 24744082
- [Background] Enard KR, Ganelin DM. Reducing preventable emergency department utilization and costs by using community health workers as patient navigators. J Healthc Manag. 2013 Nov-Dec;58(6):412-27; discussion 428. PMID 24400457
- [Background] Herman D, Conover S, Felix A, Nakagawa A, Mills D. Critical Time Intervention: an empirically supported model for preventing homelessness in high risk groups. J Prim Prev. 2007 Jul;28(3-4):295-312. doi: 10.1007/s10935-007-0099-3. Epub 2007 Jun 1. PMID 17541827
- [Background] Kangovi S, Mitra N, Grande D, Huo H, Smith RA, Long JA. Community Health Worker Support for Disadvantaged Patients With Multiple Chronic Diseases: A Randomized Clinical Trial. Am J Public Health. 2017 Oct;107(10):1660-1667. doi: 10.2105/AJPH.2017.303985. Epub 2017 Aug 17. PMID 28817334
- [Background] Kangovi S, Mitra N, Grande D, White ML, McCollum S, Sellman J, Shannon RP, Long JA. Patient-centered community health worker intervention to improve posthospital outcomes: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):535-43. doi: 10.1001/jamainternmed.2013.14327. PMID 24515422
- [Background] Kim K, Choi JS, Choi E, Nieman CL, Joo JH, Lin FR, Gitlin LN, Han HR. Effects of Community-Based Health Worker Interventions to Improve Chronic Disease Management and Care Among Vulnerable Populations: A Systematic Review. Am J Public Health. 2016 Apr;106(4):e3-e28. doi: 10.2105/AJPH.2015.302987. Epub 2016 Feb 18. PMID 26890177
- [Background] Carrasquillo O, Lebron C, Alonzo Y, Li H, Chang A, Kenya S. Effect of a Community Health Worker Intervention Among Latinos With Poorly Controlled Type 2 Diabetes: The Miami Healthy Heart Initiative Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):948-954. doi: 10.1001/jamainternmed.2017.0926. PMID 28459925
- [Background] Morgan AU, Grande DT, Carter T, Long JA, Kangovi S. Penn Center for Community Health Workers: Step-by-Step Approach to Sustain an Evidence-Based Community Health Worker Intervention at an Academic Medical Center. Am J Public Health. 2016 Nov;106(11):1958-1960. doi: 10.2105/AJPH.2016.303366. Epub 2016 Sep 15. PMID 27631747
- [Background] McBrien KA, Ivers N, Barnieh L, Bailey JJ, Lorenzetti DL, Nicholas D, Tonelli M, Hemmelgarn B, Lewanczuk R, Edwards A, Braun T, Manns B. Patient navigators for people with chronic disease: A systematic review. PLoS One. 2018 Feb 20;13(2):e0191980. doi: 10.1371/journal.pone.0191980. eCollection 2018. PMID 29462179
- [Background] Ali-Faisal SF, Colella TJ, Medina-Jaudes N, Benz Scott L. The effectiveness of patient navigation to improve healthcare utilization outcomes: A meta-analysis of randomized controlled trials. Patient Educ Couns. 2017 Mar;100(3):436-448. doi: 10.1016/j.pec.2016.10.014. Epub 2016 Oct 17. PMID 27771161
- [Background] Walkinshaw E. Patient navigators becoming the norm in Canada. CMAJ. 2011 Oct 18;183(15):E1109-10. doi: 10.1503/cmaj.109-3974. Epub 2011 Sep 19. No abstract available. PMID 21930738
- [Background] Desveaux L, McBrien K, Barnieh L, Ivers NM. Mapping variation in intervention design: a systematic review to develop a program theory for patient navigator programs. Syst Rev. 2019 Jan 8;8(1):8. doi: 10.1186/s13643-018-0920-5. PMID 30621796
- [Background] Shommu NS, Ahmed S, Rumana N, Barron GR, McBrien KA, Turin TC. What is the scope of improving immigrant and ethnic minority healthcare using community navigators: A systematic scoping review. Int J Equity Health. 2016 Jan 15;15:6. doi: 10.1186/s12939-016-0298-8. PMID 26768130